CLINICAL TRIAL: NCT01658644
Title: Put a Face to a Name (Part A): The Effects of Photographic Aids on Patient Satisfaction,Clinician Communication, and Quality of Care
Brief Title: Put a Face to a Name (Part A): The Effects of Photographic Aids on Patient Satisfaction, Clinician Communication, and Quality of Care
Acronym: Face2Name
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-0392-BE
Record Dates: First submitted 2012-08-01; First posted 2012-08-07 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2012-08

CONDITIONS: Effects of Photographic Aids (Photos of Faces) on Patient Recall of Their Clinical Care Team; Effects of Photographic Aids (Photos of Faces) on Clinician-patient Communication; Effects of Photographic Aids (Photos of Faces) on Overall Patient Satisfaction
Keywords: Patient satisfaction; Memory recall; Patient-clinician communication; health communication; clinical care team recall; hospital quality of care
MeSH Terms: conditions — Patient Satisfaction

ARMS (3):
- Group A (No Intervention): Patients participating in group A, will not be exposed to any interventions, they will partake in the typical hospital and communication experience.
- Group B (text handout) (Experimental): Patients assigned to group B will be provided with a paper or electronic version displaying a list of the names and roles of their clinical care staff; each name will NOT be accompanied by the respective photograph of each clinician. This document will be presented to the patient at the earliest possible time after admission to the hospital.
  Interventions: Other: Provision of Clinical Care Handout
- Group C (text & image handout) (Experimental): Patients assigned to group C will be provided with a paper or electronic version displaying a list of the names and roles of their clinical care staff; each name will also be accompanied by the respective photograph of each clinician. This document will be presented to the patient at the earliest possible time after admission to the hospital.
  Interventions: Other: Provision of Clinical Care Handout

INTERVENTIONS:
Other: Provision of Clinical Care Handout — Patients assigned to groups B or C will be provided with a paper or electronic version displaying either a list of the names and roles of their clinical care staff (group B), or a list of names and roles accompanied by the respective photograph of each clinician (group C). This document will be presented to the patient at the earliest possible time after admission to the hospital.
  Arms: Group B (text handout); Group C (text & image handout)

SUMMARY:
Communication is critical within healthcare, and is the root cause of most errors. With increased adoption and use of new information technologies and mediated communication systems, such as Electronic Health Records (EHR), that support visual content, hospitals can begin to look at the potential of photographic aids to improve patient satisfaction, clinician communication, and ultimately quality of care. Having pictures of clinicians and patients may improve communication by improving knowledge of who is part of the care team and may reduce electronic ordering or documentation on the wrong patient.

Despite the importance of communication between clinicians and the many advances within information and communication technologies, there is a lack of literature documenting systems that are effective at improving communication. Our research study will provide an overview on the communication models and technologies used in Canadian hospitals and add insights to the impacts of these technological adoption.

Research Question: How does the use of photographic influence patients' hospital experience?

Specifically, do photographic aids (photographs of clinicians' faces) influence:

1. Patient's ability to identify their clinical care team members
2. Patient's ability to identify their care team members and know their individual roles
3. Patient's satisfaction with their hospital experience

DETAILED DESCRIPTION:
The investigators will conduct interviews of a cross-sectional sample of patients for up to one year. There will be 2 visits during the study. The first visit should last for 15 minutes (to get consent), the second visit should last somewhere between 30 and 45 minutes. The research team created a structured survey tool designed to characterize patients' knowledge of the names and roles of their health care professionals and understanding of their plan of care, which includes some semi-structured questions to assess patient satisfaction with their hospital experience. This survey tool will be administered to participating patients each weekday during the study period, prior to their discharge from the hospital.

At the first visit, depending on whether the participant was previously assigned to group A, B or C, participants will be provided with a piece of paper listing the names of the members of their clinical care team (group B), or a piece of paper with a list of names and photographs of the members of their clinical care team (group C), or no paper at all (group A) which is currently the typical communication experience at the hospital.

There is no compensation for participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be admitted as an in-patient in the GIM ward at Toronto General Hospital.
* The ability of the patient to provide informed consent.

Exclusion Criteria:

* Patients with significant confusion, delirium or dementia will be screen by asking orientation to place and time.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Patient's memory recall of their clinical care team | up to 1 year
  Measure if there are changes in the amount of clinicians patients recognize. Measure if they are changes in the amount of clinicians' names patients can remember.

SECONDARY OUTCOMES:
Patients' satisfaction with clinician communication | up to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Appel L, Abrams H, Morra D, Wu RC. Put a face to a name: a randomized controlled trial evaluating the impact of providing clinician photographs on inpatients' recall. Am J Med. 2015 Jan;128(1):82-9. doi: 10.1016/j.amjmed.2014.08.035. Epub 2014 Sep 28. PMID 25261009